CLINICAL TRIAL: NCT06307782
Title: The Effect of Oral Whey Consumption on Insulin Resistance, Cortisol, Crp, Albumin Level
Brief Title: The Effect of Oral Whey Consumption on Insulin Resistance, Cortisol, Crp, Albumin Level and Healing Quality Before Total Hip Arthroplasty
Acronym: WHEY THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, HÜMEYRA YÜKSEL, Principal İnvestigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12833
Record Dates: First submitted 2024-01-06; First posted 2024-03-13 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-03

CONDITIONS: Crp; Insulin Resistance; Cortisol; Hypersecretion; Albus; Lichen; Quality of Life
Keywords: whey; Total Hip Arthroplasty; inflammatory; Stress; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: randomize control trials
Who Masked: Participant
Masking Description: randomize clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total Hip Arthroplasty, whey protein intake, (Experimental): In the ERAS (Enhanced Recovery After Surgery) protocol, preoperative oral carbohydrate intake must be at least 45 g. While preparing the whey mixture, 60 grams of whey powder will be mixed into 600ml bottled water to obtain a mixture worth 200 kcal. Whey will be prepared and given by the researcher at the bedside in room air using bottled water.
  In this study, by scanning the literature (13) and taking expert opinion (dietitian, anesthesiologist, orthopedic doctor), the individuals in the intervention group were given 6 hours after the surgery. It is planned to drink 600ml oral whey powder water first.
  Interventions: Dietary Supplement: whey protein intake before surgery
- Total Hip Arthroplasty, water intake (Active Comparator): 600ml of water will be given 6 hours before the surgery.
  Interventions: Dietary Supplement: Water before surgery

INTERVENTIONS:
Dietary Supplement: whey protein intake before surgery — Total Hip Arthroplasty whey protein intake,Total Hip Arthroplasty, whey protein intake,CRP,cortisol insulin resistance
  Arms: Total Hip Arthroplasty, whey protein intake,
Dietary Supplement: Water before surgery — Total Hip Arthroplasty water before surgery,Total Hip Arthroplasty, water intake,CRP,cortisol insulin resistance
  Arms: Total Hip Arthroplasty, water intake

SUMMARY:
Purpose: It was planned to determine the effect of oral whey given before total hip arthroplasty (THA) on postoperative insulin resistance, cortisol, CRP((C reactive protein), albumin level and healing quality.

Design: It was planned as Randomized Controlled. Method: Research: The study is planned to include individuals aged 50-70, who are planned for THA in the orthopedics and traumatology clinic of a public hospital, who have undergone spinal anesthesia, who have BMI <40 and ASA (American Society of Anesthesiologists)1,2,3. Individuals with endocrine or renal disorders or allergies to whey will be excluded from the study. It was planned to include at least 60 patients in the study (30 in the intervention group, 30 in the control group). It is planned to use the Patient Introduction Information Form, Physiological Measurements Chart (vital findings (blood pressure, pulse, respiratory SpO2 (pulse oximetry) value), blood glucose, cortisol, CRP and albumin value and insulin resistance) and postoperative recovery quality scale in data collection. The intervention group will be given 600 ml of oral whey 6 hours before the surgery, and the control group will be allowed to drink 600 ml of drinking water 6 hours before the surgery. 3ml of blood will be taken for blood glucose, CRP, cortisol, albumin and insulin resistance values 24 hours before the surgery, just before entering the surgery and 24 hours after the surgery. The first part of the healing quality scale is planned to be evaluated immediately before the surgery, and the second part 24 hours after the surgery.

Conclusion: When the literature was scanned, it was seen that the number of studies examining the effect of oral whey on metabolic and endocrine values in orthopedic patients was very limited and academic studies were needed. In this context, examining the effect of whey intake given before THA on the patient's blood glucose, CRP, albumin, cortisol, insulin resistance and healing quality is an original research that will contribute to the field.

DETAILED DESCRIPTION:
Total hip arthroplasty is a frequently performed and highly successful surgical intervention. It is done to relieve pain and improve function in people with advanced arthritis of the hip joint. Symptomatic osteoarthritis is the most common indication for surgery.The number of cases has increased significantly due to the rapidly increasing aging population worldwide. It is estimated that 0.33 million total hip arthroplasty (THA) are performed annually in the United States, and the demand for these surgeries will be 0.57 million in 2030. It is important to establish practical strategies to improve the quality of healthcare for patients undergoing THA and achieve earlier recovery and better outcomes, while also facilitating the reduction of the heavy economic burden associated with healthcare associated with the increased number of procedures. According to the current protocol for total hip arthroplasty, patients are kept in a fasting state from midnight to prevent the risk of pulmonary aspiration during surgery. This condition causes both physical and mental discomfort in patients. This is an old technique that has been practiced for many years. Patients experience a catabolic state after surgery, which can contribute to insulin resistance and hyperglycemia, which can worsen the stress response and prolong recovery time. Prolonged fasting in the perioperative period slows down metabolism and induces insulin resistance. Avoiding long-term fasting and metabolic satiety before surgery significantly reduces postoperative insulin resistance and also has beneficial effects on postoperative glucose and protein metabolism. Metabolic satiety prevents early feeding, preserving muscle mass and less hyperglycemia in patients. Adequate nutritional intake before and after surgery significantly reduces surgical stress and accelerates functional recovery. After whey is consumed, it passes quickly through the stomach and reaches the jejunum as intact proteins, and as clots form in the acid environment, the release of casein from the stomach is delayed. After peptic hydrolysis, peptides are released into the small intestine. It has been reported that the hydrolysis of whey in the small intestine is slow compared to other proteins, and their digestion and absorption occur over a longer intestinal length. It has been found that whey reduces food intake more at 90 minutes, but casein has a stronger effect later (at 150 minutes). It has many physiological functions, including regulating systems. However, these actions are not limited to whey proteins and peptides alone, but also result from the synergy between whey proteins and other whey components such as calcium. The effect of the proteins found in whey on satiety and food intake has an effect on the release of satiety hormones. Insulin plays a role in both short-term and long-term regulation of food intake. In the study conducted, whey plus carbohydrate drink was drunk 6 and 3 hours before surgery. Postoperative CRP (C reactive protein), albumin and insulin resistance were found to decrease significantly in those who drank whey. In a study conducted in which perioperative 2-hour fasting was administered to patients undergoing maxillofacial surgery, glutamine and oral carbohydrate solution were found to reduce postoperative insulin resistance.Whey, which will be used in this study, is easy to digest and absorb. Whey components contain significant amounts of milk proteins and their properties. The main protein of milk is casein, approximately 80% of the proteins in milk consist of whey, and the proteins in milk contain approximately 20% of the proteins. In this planned study, the effect of oral whey on postoperative surgical stress and inflammatory responses will be investigated by giving oral whey before total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 50-70,
* Spinal anesthesia
* Individuals with a BMI<40,
* Individuals with ASA I, ASA II and ASA III

Exclusion Criteria:

* Patients with communication problems
* Individuals with hepatic, renal, endocrine, gastric and neurological disorders
* Any diagnosed psychiatric disease,
* NRS (nutritional risk score )2002 score 3 Individuals with malnutrition and above,
* Allergy to whey and lactose intolerance will be excluded from the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of C Reactive Protein | 24 hour
  physiological parameter, questionnaire
Rate of insulin resistance | 24 hour
  physiological parameter, questionnaire
Rate of albumen | 24 hour
  physiological parameter, questionnaire
Rate of cortisol | 24 hour
  physiological parameter, questionnaire
Healing Quality | 24 hour
  Quality of Recovery-15 scala

CONTACTS AND LOCATIONS:
Locations (1):
- HÜMEYRA, Nevşehir, Nevşehir Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
randomize clinical study

REFERENCES:
- [Background] 1.Ferguson R, Palmer A, Taylor A, Porter M, Malchau H, Jones S,G(2018). Hip replacement. Lancet.392(10158):1662-1671 2.Kurtz S, Ong K, Lau E, Mowat F, Halpern M(2007). 2005'ten 2030'a kadar Amerika Birleşik Devletleri'nde primer ve revizyon kalça ve diz artroplastisinin projeksiyonları. J Bone Joint Surg Am; 89 :780-785. 3. Kaye A, Urman R, Cornett E, Hart B, Chami A, Gayle J, et al(2019). Ortopedik cerrahide geliştirilmiş iyileşme yolları. J Anesteziol Clin Pharmacol.; 35 :35-39. 4. Kehlet H(1997). Postoperatif patofizyoloji ve rehabilitasyonu kontrol etmek için multimodal yaklaşım. Br J Anaesth.; 78 :606-617. 5.Nygren J (2006). The metabolic effects of fasting and surgery. Best Practice & Research Clinical Anaesthesiology.20(3):429-438 6. Luhovyy BL, Akhavan T, Anderson GH. Whey proteins in the regulation of food intake and satiety. J Am Coll Nutr. 2007;26(6):704S-12S. doi:10.1080/07315724.2007.10719651 7. Zemel MB. Mechanisms of dairy modulation of adiposity. J. Nutr.2003;133:252S-256S 8. Perrone F, da-Silva-Filho AC, Adôrno IF, Anabuki NT, LealFS, Colombo T, da Silva BD, Dock-Nascimento DB, Damiao A, da Aguilar-Nascimento JE(2011). Effects ofpreoperative feeding with a whey protein plus carbohydrate drink on the acute phase response and insulin resistance. A randomized trial. Nutr J.;10:66. 9. Singh M, Chaudhary M, Vashistha A, Kaur G (2015). Evaluation of effects of a preoperative 2-hour fast with glutamine and carbohydrate rich drink on insulin resistance in maxillofacial surgery. J Oral Biol Craniofac Res.5(1):34-9 10. Güzeler N, Esmek E,M, & Kalender M (2017). Peyniraltı Suyu ve Peyniraltı Suyunun İçecek Sektöründe Değerlendirilme Olanakları. Çukurova Tarım Gıda Bil. Der.32(2);27-36